CLINICAL TRIAL: NCT00128557
Title: A Randomized Community Trial of Newborn Vitamin A Supplementation to Reduce Infant Mortality in Rural Bangladesh
Brief Title: Community Trial of Newborn Vitamin A Supplementation to Reduce Infant Mortality in Rural Bangladesh
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Johns Hopkins University (Other); Bill and Melinda Gates Foundation (Other); Canadian International Development Agency (Other Government); Access Business Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: H.22.03.01.09.A2
Record Dates: First submitted 2005-08-09; First posted 2005-08-10 (Estimated); Last update posted 2022-10-03 (Actual); Status verified 2007-04

CONDITIONS: Mortality Through Six Months of Age; Vitamin A Deficiency
Keywords: Vitamin A; Newborn health; Infant Mortality; Supplementation; Micronutrients; Bangladesh
MeSH Terms: conditions — Vitamin A Deficiency; Infant Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Supplement containing soybean oil with a small amount of vitamin E as an antioxidant
  Interventions: Dietary Supplement: vitamin A supplementation (15,000 ug retinol equivalents or 50,000 IU)
- Vitamin A (Active Comparator): 15,000 ug retinol equivalents (50,000 International Units)
  Interventions: Dietary Supplement: vitamin A supplementation (15,000 ug retinol equivalents or 50,000 IU)

INTERVENTIONS:
Dietary Supplement: vitamin A supplementation (15,000 ug retinol equivalents or 50,000 IU) — Single dose of 15,000 ug retinol equivalents at or near birth vs a placebo

SUMMARY:
The purpose of this trial is determine whether a 50,000 IU oral dose of vitamin A delivered to newborn infants within the first days of life, reduces six-month infant mortality by at least 15%. The trial will also evaluate whether the survival impact of newborn vitamin A dosing is modified by concurrent weekly, routine maternal vitamin A or beta-carotene supplementation during pregnancy through three months postpartum, gestational age and birth size.

DETAILED DESCRIPTION:
This is a randomized, double-masked, placebo-controlled, community trial of newborn vitamin A supplementation on mortality in the first six months of life. The trial is being implemented in 596 sectors (i.e. villages and/or smaller groupings), in two thanas comprising a population of ~580,000 in rural northern Bangladesh (Gaibandha/Rangpur area) and is nested within the JiVitA-1 maternal supplementation study. Women residing in the study area are already under 5-weekly pregnancy surveillance conducted by village-based field staff as part of the maternal supplementation trial. During their third trimester of pregnancy, women are visited by a study supervisor who explains the purpose and procedures of the study. After obtaining informed consent, women are interviewed for possible risk factors in the third trimester of pregnancy, including a 30-day history of morbidity, a 7-day dietary and alcohol intake and tobacco use questionnaire, a 7-day household chores questionnaire, and maternal anthropometry (mid upper arm circumference measurement). Upon birth, household members contact the village-based field staff who immediately administers the vitamin A or placebo to the infant, according to sector assignment. After supplementation, newborns are measured for weight, length and mid-upper arm, head and chest circumference, and then followed weekly for vital status for three months, and again at six months of age. A child death initiates the process of death verification and cause of death determination.

ELIGIBILITY:
Inclusion Criteria: Infants born to women enrolled in a maternal supplementation trial, alive and less than 30 days of age during a newborn dosing visit Exclusion Criteria: Infants who died before the dose could be administered or infants older than 30 days at the time of dosing

Ages: 1 Minute to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15937 (Actual)
Dates: Start 2004-01; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
24-week infant mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Rolf DW Klemm, Dr PH, Principal Investigator — Johns Hopkins University; Keith P West, Jr., Dr. P.H., Study Director — Johns Hopkins Bloomberg School of Public Health; Parul Christian, Dr. P.H., Study Director — Johns Hopkins Bloomberg School of Public Health; Mahbubar Rashid, MBBS, MSc, MBA, Study Director — JiVitA Bangladesh Project; Alain B. Labrique, MSc, Study Director — Johns Hopkins Bloomberg School of Public Health; Alfred Sommer, M.D., Study Director — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- JiVitA Bangladesh Project, Rangpur, Rajshahi Division, Bangladesh

REFERENCES:
- [Derived] Ali H, Hamadani J, Mehra S, Tofail F, Hasan MI, Shaikh S, Shamim AA, Wu LS, West KP Jr, Christian P. Effect of maternal antenatal and newborn supplementation with vitamin A on cognitive development of school-aged children in rural Bangladesh: a follow-up of a placebo-controlled, randomized trial. Am J Clin Nutr. 2017 Jul;106(1):77-87. doi: 10.3945/ajcn.116.134478. Epub 2017 May 10. PMID 28490513
- [Derived] Coles CL, Labrique A, Saha SK, Ali H, Al-Emran H, Rashid M, Christian P, West KP Jr, Klemm R. Newborn vitamin A supplementation does not affect nasopharyngeal carriage of Streptococcus pneumoniae in Bangladeshi infants at age 3 months. J Nutr. 2011 Oct;141(10):1907-11. doi: 10.3945/jn.111.141622. Epub 2011 Aug 10. PMID 21832026